CLINICAL TRIAL: NCT00216385
Title: A Randomised Open-Label Controlled Trial of a 4-Month Gatifloxacin-Containing Regimen Versus Standard Regimen for the Treatment of Adult Patients With Pulmonary Tuberculosis
Brief Title: A Controlled Trial of a 4-Month Quinolone-Containing Regimen for the Treatment of Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: World Health Organization (Other); European Commission (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICA4-CT 2002-10057
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Treatment; Quinolone; Short course chemotherapy
MeSH Terms: conditions — Tuberculosis

INTERVENTIONS:
Drug: Gatifloxacin combined regimen

SUMMARY:
Tuberculosis is currently treated with a 6-month course regimen. During this time many patients might fail to adhere to treatment and default, increasing the risk of recurrent disease which might be multidrug resistant. A shorter duration of treatment is expected to provide improved patient compliance and at least equal or better clinical outcome. The aim of the trial is to evaluate the efficacy and safety of a gatifloxacin-containing regimen of four months duration for the treatment of pulmonary tuberculosis,

DETAILED DESCRIPTION:
In order to evaluate the efficacy and safety of the 4-month test gatifloxacin-containing regimen, comparison will be made with a standard 6-month regimen, recommended by WHO. Patients will be treated with one of the two regimens that will be randomly allocated. A total of 2070 patients will ne recruited in the trial and followed-up for a duration of 2 years. The trial is multicentre, and conducted in 5 countries in Africa.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Aged 18 to 65 years
* Currently suffering from recently diagnosed microscopically proven pulmonary tuberculosis and providing informed consent for inclusion in the study.

Exclusion Criteria:

* Patients with history of tuberculosis treatment within the last 3 years
* History of diabetes mellitus or non insulin dependent diabetes mellitus requiring treatment
* Concomitant infection requiring additional anti-infective treatment (especially anti-retroviral therapy)
* HIV infected patients with WHO stage 3 infection - except those presenting with only the "loss of weight>10% body weight" criterion - and all HIV infected patients at WHO stage 4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2070
Dates: Start 2005-01; Study Completion 2008-12

PRIMARY OUTCOMES:
Efficacy: Percentage of relapses by 24 months following treatment cure
Safety: Percentage of adverse events

SECONDARY OUTCOMES:
Efficacy: Time to relapse
Efficacy: Percentage of smear and culture conversion at 8 weeks
Efficacy: Percentage of patient cured at the end of treatment
Efficacy: Time to a composite "unsatisfactory" endpoint
Safety outcome: Distribution of type and grading of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lienhardt, MD, Study Director — Institut de Recherche pour le Developpement
Locations (5):
- Programme National de Lutte contre la Tuberculose, Cotonou, Benin
- Service Pneumo-Phtisiologie, CHU Ignace Deen, Conakry, Guinea
- Kenya Medical Research Institute, Nairobi, Kenya
- Programme National de Lutte contre la Tuberculose, Dakar, Senegal
- Medical Research Council, Durban, KwaZulu, South Africa

REFERENCES:
- [Derived] Pasipanodya JG, Smythe W, Merle CS, Olliaro PL, Deshpande D, Magombedze G, McIlleron H, Gumbo T. Artificial intelligence-derived 3-Way Concentration-dependent Antagonism of Gatifloxacin, Pyrazinamide, and Rifampicin During Treatment of Pulmonary Tuberculosis. Clin Infect Dis. 2018 Nov 28;67(suppl_3):S284-S292. doi: 10.1093/cid/ciy610. PMID 30496458
- [Derived] Olliaro PL, Merle C, Mthiyane T, Bah B, Kassa F, Amukoye E, N Diaye A, Perronne C, Lienhardt C, McIlleron H, Fielding K. Effects on the QT Interval of a Gatifloxacin-Containing Regimen versus Standard Treatment of Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2017 Jun 27;61(7):e01834-16. doi: 10.1128/AAC.01834-16. Print 2017 Jul. PMID 28438924
- [Derived] Merle CS, Fielding K, Sow OB, Gninafon M, Lo MB, Mthiyane T, Odhiambo J, Amukoye E, Bah B, Kassa F, N'Diaye A, Rustomjee R, de Jong BC, Horton J, Perronne C, Sismanidis C, Lapujade O, Olliaro PL, Lienhardt C; OFLOTUB/Gatifloxacin for Tuberculosis Project. A four-month gatifloxacin-containing regimen for treating tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1588-98. doi: 10.1056/NEJMoa1315817. PMID 25337748
- [Derived] Smythe W, Merle CS, Rustomjee R, Gninafon M, Lo MB, Bah-Sow O, Olliaro PL, Lienhardt C, Horton J, Smith P, McIlleron H, Simonsson US. Evaluation of initial and steady-state gatifloxacin pharmacokinetics and dose in pulmonary tuberculosis patients by using monte carlo simulations. Antimicrob Agents Chemother. 2013 Sep;57(9):4164-71. doi: 10.1128/AAC.00479-13. Epub 2013 Jun 17. PMID 23774436
- [Derived] Merle CS, Sismanidis C, Sow OB, Gninafon M, Horton J, Lapujade O, Lo MB, Mitchinson DA, Perronne C, Portaels F, Odhiambo J, Olliaro P, Rustomjee R, Lienhardt C, Fielding K. A pivotal registration phase III, multicenter, randomized tuberculosis controlled trial: design issues and lessons learnt from the Gatifloxacin for TB (OFLOTUB) project. Trials. 2012 May 18;13:61. doi: 10.1186/1745-6215-13-61. PMID 22607233